CLINICAL TRIAL: NCT03494335
Title: Online Surveys to Assess the Perception and Performance of Imaging Associated Aspects
Brief Title: Online Surveys to Assess the Perception and Performance of Imaging and Associated Aspects
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled.
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Michael V Knopp MD PhD, Professor, University of Cincinnati
Other Study IDs: RP0320_S02/2018E0141
Record Dates: First submitted 2018-03-30; First posted 2018-04-11 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Perception of Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Volunteer participants: Volunteer participants will participate in surveys assessing their perception of various imaging aspects.
  Interventions: Other: Online surveys

INTERVENTIONS:
Other: Online surveys — The investigators are recruiting health care providers for these surveys that are involved in or use imaging.

SUMMARY:
In this exploratory study, the researchers would like to investigate the background, perception, current use practices, potential unmet needs and/or challenges in regard to imaging procedures, imaging technology, or any other aspect related to the broader field of imaging.

DETAILED DESCRIPTION:
The researchers plan to include volunteer participants to complete these surveys. The goal of these exploratory efforts will be to increase the currently very limited information available in the topics of interest stated above, and the findings, even if only from limited group of respondents, will help guide research development, prepare for design of clinical trials, guide special interest groups, and serve as role data for appropriate scientific publications.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who have access to the online survey tool and can read and write in English

Exclusion Criteria:

* None, as this is voluntary

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of volunteers agreeing to complete the survey tool. It is anticipated that the surveys will be completed by participants that can be considered stakeholders, such as physicians, technologist's physicists, imaging scientists, administrative staff, or others with interest in the topic.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-08-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Perception of PET/CT imaging agent Y-90 | through study completion, on average 2-5 years
  To evaluate participants' perceptions of Y-90 using a likert scale on an online survey
Perception of PET/CT imaging agent NaF | through study completion, on average 2-5 years
  To evaluate participants' perceptions of NaF using a likert scale on an online survey
Perception of MRI contrast agents | through study completion, on average 2-5 years
  To evaluate participants' perceptions of MR contrast agents using a likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Michael V Knopp, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- Martha Morehouse Medical Plaza, Columbus, Ohio, United States

DOCUMENTS (1):
  • Study Protocol (2017-10-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT03494335/Prot_000.pdf